CLINICAL TRIAL: NCT01247675
Title: A Phase 2, Multiple Dose, Open-Label, Parallel-Group, Active Controlled, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of ACP-001 in Adult Patients With Growth Hormone Deficiency
Brief Title: A Safety, Pharmacokinetic and Pharmacodynamic Study of ACP-001 (TransCon hGH) in Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACP-001 CT-002
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ACP-001, 0.02 mg hGH/kg/wk (Experimental): Once weekly subcutaneous injection of ACP-001 equivalent to 0.02 mg hGH/kg/week for 4 weeks
  Interventions: Drug: ACP-001 (TransCon hGH)
- ACP-001, 0.04 mg hGH/kg/wk (Experimental): Once weekly subcutaneous injection of ACP-001 equivalent to 0.04 mg hGH/kg/week for 4 weeks
  Interventions: Drug: ACP-001 (TransCon hGH)
- ACP-001, 0.08 mg hGH/kg/wk (Experimental): Once weekly subcutaneous injection of ACP-001 equivalent to 0.08 mg hGH/kg/week for 4 weeks
  Interventions: Drug: ACP-001 (TransCon hGH)
- Omnitrope, 0.04 mg hGH/kg/wk (Active Comparator): Once daily subcutaneous injection of human Growth Hormone (Omnitrope) equivalent to 0.04 mg hGH/kg/week for 4 weeks
  Interventions: Drug: Omnitrope

INTERVENTIONS:
Drug: ACP-001 (TransCon hGH) — s.c., weekly injection
  Arms: ACP-001, 0.02 mg hGH/kg/wk
Drug: ACP-001 (TransCon hGH) — s.c., weekly injection
  Arms: ACP-001, 0.04 mg hGH/kg/wk
Drug: ACP-001 (TransCon hGH) — s.c., weekly injection
  Arms: ACP-001, 0.08 mg hGH/kg/wk
Drug: Omnitrope — s.c., daily injection
  Arms: Omnitrope, 0.04 mg hGH/kg/wk

SUMMARY:
This study investigates the safety, tolerability, pharmacokinetic profile (PK), and pharmacodynamic response (PD) of three different doses of ACP-001 given once-a-week compared to one dose-level of an approved daily human growth hormone product over a period of 4 weeks (4 weekly administrations versus 28 daily administrations) in adults with Growth Hormone Deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 20 to 70 years
* Body Mass Index (BMI, kg/m2) of 19.0 to 36.0 kg/m2, both inclusive
* Adult Growth Hormone Deficient (AHGD) patients with documented growth hormone deficiency as defined in the Consensus guidelines for the diagnosis and treatment of adults with GH deficiency II (Consensus Guidelines 1998 and 2007)
* Fertile females must agree to use appropriate contraceptive methods and have a negative pregnancy test at inclusion
* GH replacement therapy for at least 3 months
* Willing to maintain current activity level during the trial
* Subjects are able and willing to provide written informed consent and authorization for protected health information disclosure in accordance with Good Clinical Practice (GCP)

Exclusion Criteria:

* History of hypersensitivity and/or idiosyncrasy to any of the test compounds or excipients employed in this study.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods. Reliable methods for women are orally administered hormonal contraceptives, surgical intervention (e.g. tubal ligation), intrauterine device (IUD) and sexual abstinence.
* Active malignant disease or malignant disease within the last 5 years
* Proliferative retinopathy judged by retina-photo within the last year
* Heart insufficiency as judged by the investigator and/or NYHA 3 or greater (NYHA criteria for diagnosis of diseases of the heart, 1994)
* Subjects with uncontrolled diabetes with an HbA1c above 8.0% and/or insulin treatment
* Stable pituitary hormone replacement therapy for less than 3 months
* Impaired liver function as judged by the investigator or hepatic transaminases > 2 times the upper limit of normal
* Impaired kidney function as judged by the investigator and/or creatinine clearance <50 mL/min and/or serum creatinine > 1.4 mg/dL
* Participation in another interventional clinical study involving an investigational compound within 3 months prior to enrolment in this study or participation in another interventional clinical study involving an investigational compound during this study.
* Subjects who are unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study.
* History or presence of alcohol abuse or drug abuse.
* Patients with known history for, or presence of, anti-hGH and / or anti-PEG antibodies

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beckert, MD, Study Director — Ascendis Pharma A/S
Locations (4):
- Aarhus University Hospital, Aarhus, Denmark
- Charité University Hospital Berlin, Berlin, Germany
- University Hospital Genova, Genova, Italy
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ACP-001, 0.02 mg hGH/kg/wk: ACP-001 (TransCon hGH): subcutaneous, weekly injection equivalent to 0.02 mg hGH/kg/wk over 4 weeks. Prior to randomization, study subjects entered a 14 to 21 day wash out period following cessation of daily growth hormone therapy.
- ACP-001, 0.04 mg hGH/kg/wk: ACP-001 (TransCon hGH): subcutaneous, weekly injection equivalent to 0.04 mg hGH/kg/wk over 4 weeks. Prior to randomization, study subjects entered a 14 to 21 day wash out period following cessation of daily growth hormone therapy.
- ACP-001, 0.08 mg hGH/kg/wk: ACP-001 (TransCon hGH): subcutaneous, weekly injection equivalent to 0.08 mg hGH/kg/wk over 4 weeks. Prior to randomization, study subjects entered a 14 to 21 day wash out period following cessation of daily growth hormone therapy.
- Omnitrope, 0.04 mg hGH/kg/wk: Human Growth Hormone: subcutaneous, daily injection of Omnitrope equivalent to 0.04 mg/kg/wk over 4 weeks. Prior to randomization, study subjects entered a wash out period of 14 to 21 days following cessation of daily growth hormone therapy.
Period: Overall Study
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
Started | 10 | 10 | 9 | 8
Completed | 8 | 8 | 9 | 8
Not Completed | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACP-001, 0.02 mg hGH/kg/wk: ACP-001 (TransCon hGH): s.c., weekly injection equivalent to 0.02 mg hGH/kg/wk for 4 weeks
- ACP-001, 0.04 mg hGH/kg/wk: ACP-001 (TransCon hGH): s.c., weekly injection equivalent to 0.04 mg hGH/kg/wk for 4 weeks
- ACP-001, 0.08 mg hGH/kg/wk: ACP-001 (TransCon hGH): s.c., weekly injection equivalent to 0.08 mg hGH/kg/wk for 4 weeks
- Omnitrope, 0.04 mg hGH/kg/wk: Human Growth Hormone: s.c., daily injection equivalent to 0.04 mg hGH/kg/wk for 4 weeks
- Total: Total of all reporting groups
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk | Total
Number analyzed (Participants) | 10 | 10 | 9 | 8 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.6) | 45.9 (15.0) | 51.6 (18.1) | 44.0 (15.7) | 49.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 3 | 19
  Male | 5 | 4 | 4 | 5 | 18
Weight [Mean (Standard Deviation); unit: kg] | 82.3 (19.8) | 79.6 (17.0) | 92.5 (20.5) | 74.7 (16.6) | 82.4 (18.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 27.6 (4.4) | 27.9 (4.4) | 30.7 (4.4) | 25.7 (4.4) | 28.0 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Tolerability Events (Assessed by the Patient and Investigator)
Description: Assessment of local tolerability was performed by examining injection sites by the investigator during study visits, and on the basis of records in the Patient Diary. Assessments included erythema, swelling, or pain.
Time Frame: Start of study treatment through Week 4
Population: All patients who were randomized and received at least one dose of test product were included in the Safety analysis.
Measure: Number; unit: Number of subjects with any symptom
Groups:
- Omnitrope, 0.04 mg hGH/kg/wk: Human Growth Hormone: s.c., daily injection of Omnitrope equivalent to 0.04 mg hGH/kg/wk for 4 weeks
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
Number analyzed (Participants) | 10 | 10 | 9 | 8
Number of subjects with any symptom | 3 | 3 | 2 | 1

2. Primary Outcome: Incidence of Treatment Emergent Anti-hGH Binding Antibody Formation
Description: Number of subjects with treatment emergent anti-hGH binding antibodies
Time Frame: Start of study treatment through Day 42
Population: All patients who were randomized and received at least one dose of test product were included in the Safety analysis.
Measure: Number; unit: Participants
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
Number analyzed (Participants) | 10 | 10 | 9 | 8
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Cmax of hGH
Description: As part of the following endpoint:
  Pharmacokinetic (PK) profile of serum human Growth Hormone (hGH) from ACP-001 treated dose groups compared to the PK profile of hGH from the daily Omnitrope treated group.
  Cmax (maximum value of concentration) values at Week 4
Time Frame: Days 22 to 29
Population: Pharmacokinetic and pharmacodynamic analysis was performed on all patients who had at least one measurement of the primary variable and who had attended the Day 28 study visit. Two patients in Cohort 2 (ACP-001, 0.04 mg hGH/kg/wk) were withdrawn from the study before Day 28 and were therefore excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
Number analyzed (Participants) | 10 | 8 | 9 | 8
ng/mL | 1.2 (0.8) | 1.9 (0.9) | 3.8 (2.0) | 2.0 (1.1)

4. Secondary Outcome: Emax of IGF-I
Description: As part of the following endpoint:
  Pharmacodynamic (PD) response of serum Insulin-like Growth Factor-I (IGF-I) from ACP-001 treated dose groups compared to the PD response of IGF-I from the daily Omnitrope treated group.
  Emax (maximum observed response) values at Week 4
Time Frame: Days 22 to 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ACP-001, 0.04 mg hGH/kg/wk: ACP-001 (TransCon hGH): s.c., weekly injection equivalent to 0.04 mg hGH/kg/wk
- ACP-001, 0.08 mg hGH/kg/wk: ACP-001 (TransCon hGH): s.c., weekly injection equivalent to 0.08 mg hGH/kg/wk
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
Number analyzed (Participants) | 10 | 8 | 9 | 8
ng/mL | 71.8 (26.9) | 108.6 (91.7) | 125.6 (70.1) | 109.8 (37.1)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events include events starting on or after Day 0 and ending on or before Day 42.
Description: A subject with more than one finding in a specific category was only counted once.
Arm/Group | ACP-001, 0.02 mg hGH/kg/wk | ACP-001, 0.04 mg hGH/kg/wk | ACP-001, 0.08 mg hGH/kg/wk | Omnitrope, 0.04 mg hGH/kg/wk
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 6/10 | 9/10 | 7/9 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-001, 0.02 mg hGH/kg/wk (N=10) | ACP-001, 0.04 mg hGH/kg/wk (N=10) | ACP-001, 0.08 mg hGH/kg/wk (N=9) | Omnitrope, 0.04 mg hGH/kg/wk (N=8)
Severe Adrenal Crisis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient had a history of adrenal crisis
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-001, 0.02 mg hGH/kg/wk (N=10) | ACP-001, 0.04 mg hGH/kg/wk (N=10) | ACP-001, 0.08 mg hGH/kg/wk (N=9) | Omnitrope, 0.04 mg hGH/kg/wk (N=8)
Fatigue (General disorders) | 3 (8) | 3 (4) | 1 (4) | 2 (12)
Application site erythema (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Application site induration (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Application site pruritus (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 1 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (7) | 2 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Affect lability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other